CLINICAL TRIAL: NCT07340528
Title: Endoscopically Assisted Management of Maxillofacial Fractures: A Prospective Study on Efficacy and Outcomes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Elhossieny abdelaal mohamed, principal investigator, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med--25-12-4Md
Record Dates: First submitted 2026-01-04; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Maxillofacial Injuries; Maxillofacial Trauma; Subcondylar Process of Mandible Closed Fracture; Orbital Floor (Blow-Out) Closed Fracture; Frontal Sinus Fracture
Keywords: maxillofacial; fractures; endoscopic
MeSH Terms: conditions — Maxillofacial Injuries; Fractures, Closed; Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- endoscopic assisted reduction and fixation of maxillofacial fractures (Other)
  Interventions: Procedure: endoscopy assisted management of maxillofacial fractures

INTERVENTIONS:
Procedure: endoscopy assisted management of maxillofacial fractures — using small hidden incisions to approach fractures instead of direct classic approaches

SUMMARY:
The goal of this clinical trial is to assess the efficacy of endoscopically assisted management of maxillofacial fractures in terms of fracture reduction, stability, and functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

Patients with the following maxillofacial fractures (zygomaticomaxillary complex, orbital floor, mandibular condyle and frontal sinus fracture)

Exclusion Criteria:

* Patients with Severe comminuted fractures requiring extensive open reconstruction
* Patients unfit for intervention medically

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2028-01-15 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
rate of facial nerve injury | day 1

SECONDARY OUTCOMES:
operating time | periprocedural

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 20 years

REFERENCES:
- [Background] Pham AM, Strong EB. Endoscopic management of facial fractures. Curr Opin Otolaryngol Head Neck Surg. 2006 Aug;14(4):234-41. doi: 10.1097/01.moo.0000233593.84175.6e. PMID 16832179
- See also: Related Info — https://journals.lww.com/co-otolaryngology/abstract/2006/08000/endoscopic_management_of_facial_fractures.3.aspx